CLINICAL TRIAL: NCT06770218
Title: Effects of Pelvic Girdle Stability Training With and Without Therapeutic Taping on Trunk Control in Childern With Down Syndrome
Brief Title: Effects of Pelvic Girdle Stabililty With Use of Therapeutic Taping in Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0713
Record Dates: First submitted 2024-11-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome
Keywords: Down syndrome; therapeutic taping; trunk control; pelvic girdle
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: it will be randomized contrail in which non probability convenient sampling will be used two groups of A and B .Group A will given therapeutic training nd B group pelvic girdle training without therapeutic training
Who Masked: Participant
Masking Description: single participatnts will get seperate treatment protocols and possible efforts will b put to make the both groups about ther treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): A 8 groups individuals will receive pelvic girdle stability training along with therapeutic taping.
  Interventions: Other: pelvic girdle stability training and therapeutic tapping
- control group (Other): pelvic stability through targeted exercises without the inclusion of therapeutic taping exercise including pelvic bridge, one leg bridge
  Interventions: Other: pelvic girdle stability training only

INTERVENTIONS:
Other: pelvic girdle stability training and therapeutic tapping — pelvic girdle stability training performed along with therapeutic taping in experimental group tapping involves applying strips one and two over the paraspinal region from l4 to t1 in a caudo cephalic directions. strips 3 and 4 along the lower portion of trapezius with a medially directed force from the acromion process to T12 obliquely. total session time 45 minutes to 60 minutes
  Arms: experimental group
Other: pelvic girdle stability training only — participates engaged in pelvic girdle stability training focusing on exercises therapeutics taping was not be administrated during these stability exercises. excercise include pelvic brigde, one leg bridge, calm exercise for gluteus medius, leg lift 4 point kneelig arm lift
  Arms: control group

SUMMARY:
A Interventional study on 16 down syndrome pateints and check effects o therapeutic taping on pelvic girdle stability on 8 weeks sessions

DETAILED DESCRIPTION:
Study group A will undergo pelvic girdle stablilty traing along with therapeutic taping and group B will receive pelvic girdle satbility traing of 8 weeks and chcek the effects by trunk control assessement tool,gross motor functional scale .this study type is conviennet sampling techniques and check effetcts by exercising

ELIGIBILITY:
Inclusion Criteria:

* Functional hearing and vision
* Ability to understand commands.

Exclusion Criteria:

* Children with severe mental retardation
* History of trauma and surgery'

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
trunk control assesment scale | 6 weeks
  a tool having 58 points. 20 points cooresponds to static balance and 28 for selective movement control other 10 point for dynamic reaching.

SECONDARY OUTCOMES:
GMFCS-88 | 6 weeks
  A Tool use for gross motor functional level having 88 points will use before and after application of taping.

CONTACTS AND LOCATIONS:
Overall Officials: Maham Javed, MS*, Principal Investigator — Ripah International university
Locations (2):
- Pakistan (2):
  - Riphah international university. lahore pakistan., Lahore, Punjab Province
  - Riphah international university, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giustino V, Messina G, Alesi M, La Mantia L, Palma A, Battaglia G. Study of posturalcontrol and body balance in subjects with Down syndrome. Human Movement. 2021;22(1):66-71.